CLINICAL TRIAL: NCT06172439
Title: The Effect Of Acupressure Applıcatıon On Postoperative Pain Level İn Women With Abdominal Gynecologıcal Surgery: Randomized Controlled Study
Brief Title: Effect of Acupressure on Postoperative Pain With Gynecologıcal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Meliha Dönmez, master student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBU-MDONMEZ-001
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Acupressure; Post Operative Pain; Nurse's Role
MeSH Terms: conditions — Pain, Postoperative | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled intervention trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Women in the intervention group will receive acupressure for 12 minutes.
  Interventions: Other: acupressure
- control group (No Intervention): Women in the control group will not receive acupressure and will continue with routine care.

INTERVENTIONS:
Other: acupressure — Women in the intervention group will receive acupressure for 12 minutes.The acupressure pressure points related to the gynecologic surgery to be performed are named as the large intestine (LI4), stomach (ST36) and spleen (SP6) meridians, respectively. These points are determined by expert opinion and are used for pain control.
  Arms: experimental group

SUMMARY:
In this study, the effect of acupressure on postoperative pain level in women with abdominal gynecologıcal surgery will be studied and it will be conducted as a randomized controlled intervention study to examine the relationships with each other.The sample group will consist of 102 women, 51 in the intervention group and 51 in the control group.Within the scope of the study, the data will be collected using the 'Personal Information Form and Short-Form McGill Pain Questionnaire (SF-MPQ)' created by the researcher. Data will be analyzed using SPSS-26 package.

DETAILED DESCRIPTION:
In this study, the effect of acupressure on postoperative pain level in women with abdominal gynecologıcal surgery will be studied and it will be conducted as a randomized controlled intervention study to examine the relationships with each other.The sample group will consist of 102 women, 51 in the intervention group and 51 in the control group.Within the scope of the study, the data will be collected using the 'Personal Information Form and Short-Form McGill Pain Questionnaire(SF-MPQ)' created by the researcher. Data will be obtained by the researcher by faceto-face interviews with women. In addition, women in the intervention group will receive acupressure once on postoperative days 0 and 1. Acupressure points related to gynecological surgery (large intestine (LI4), stomach (ST36) and spleen (SP6)) will be applied for a total of 12 minutes with 2 minutes of pressure on each point. Women in the control group will continue their routine care. Data will be evaluated with SPSS-26 package.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older,
* Being literate,
* To be able to understand and speak Turkish,
* No deformity or lesion in the areas where acupressure will be applied,
* Undergoing abdominal gynecologic surgery with general anesthesia,
* Any narcotic or epidural for pain control after surgery lack of analgesia
* Participation in the routine pain protocol of the clinic

Exclusion Criteria:

* The presence of any systemic disease that causes chronic pain,
* Receiving spinal or epidural anesthesia,
* Patients who are administered narcotic or any analgesic drug other than the routine pain protocol applied in the clinic after surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
postoperative pain level | 7 month
  Pain will be measured with the Short-Form McGill pain questionnaire (SF-MPQ) before and after the application

CONTACTS AND LOCATIONS:
Overall Officials: Meliha Dönmez, Principal Investigator — Saglik Bilimleri Universitesi; Gülşah Kök, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Faculty of nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kidanemariam BY, Elsholz T, Simel LL, Tesfamariam EH, Andemeskel YM. Utilization of non-pharmacological methods and the perceived barriers for adult postoperative pain management by the nurses at selected National Hospitals in Asmara, Eritrea. BMC Nurs. 2020 Oct 22;19:100. doi: 10.1186/s12912-020-00492-0. eCollection 2020. PMID 33110397
- [Background] Bernardinelli N, Valery A, Barrault D, Dorland JM, Palut P, Toumi H, Lespessailles E. Effectiveness of Shiatsu on Fatigue in Patients with Axial Spondyloarthritis: Protocol for a Randomized Cross-Over Pilot Study. Rheumatol Ther. 2023 Aug;10(4):1107-1117. doi: 10.1007/s40744-023-00558-w. Epub 2023 May 12. PMID 37173568
- [Background] Mehta P, Dhapte V, Kadam S, Dhapte V. Contemporary acupressure therapy: Adroit cure for painless recovery of therapeutic ailments. J Tradit Complement Med. 2016 Jul 22;7(2):251-263. doi: 10.1016/j.jtcme.2016.06.004. eCollection 2017 Apr. PMID 28417094
- [Background] Borys M, Zyzak K, Hanych A, Domagala M, Galkin P, Galaszkiewicz K, Klaput A, Wroblewski K, Miekina J, Onichimowski D, Czuczwar M. Survey of postoperative pain control in different types of hospitals: a multicenter observational study. BMC Anesthesiol. 2018 Jul 18;18(1):83. doi: 10.1186/s12871-018-0551-3. PMID 30021520
- [Background] Erden S, Guler S, Tura I, Basibuyuk IF, Arslan UE. Evaluating patient outcomes in postoperative pain management according to the revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R). Appl Nurs Res. 2023 Oct;73:151734. doi: 10.1016/j.apnr.2023.151734. Epub 2023 Aug 18. PMID 37722782
- [Background] Mohd Nafiah NA, Chieng WK, Zainuddin AA, Chew KT, Kalok A, Abu MA, Ng BK, Mohamed Ismail NA, Nur Azurah AG. Effect of Acupressure at P6 on Nausea and Vomiting in Women with Hyperemesis Gravidarum: A Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Sep 1;19(17):10886. doi: 10.3390/ijerph191710886. PMID 36078602
- [Background] Noll E, Shodhan S, Romeiser JL, Madariaga MC, Page C, Santangelo D, Guo X, Pryor AD, Gan TJ, Bennett-Guerrero E. Efficacy of acupressure on quality of recovery after surgery: Randomised controlled trial. Eur J Anaesthesiol. 2019 Aug;36(8):557-565. doi: 10.1097/EJA.0000000000001001. PMID 30985537
- [Background] Alimoradi Z, Kazemi F, Valiani M, Gorji M. Comparing the effect of auricular acupressure and body acupressure on pain and duration of the first stage of labor: study protocol for a randomized controlled trial. Trials. 2019 Dec 23;20(1):766. doi: 10.1186/s13063-019-3896-0. PMID 31870458